CLINICAL TRIAL: NCT03483636
Title: Single-Center, Double-Blind, Placebo-Controlled, Single-Dose, 4-Period Crossover, Drug-Alcohol Interaction Study in Lemborexant in Healthy Subjects
Brief Title: Study of Lemborexant-Alcohol Interaction in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: E2006-A001-009
Record Dates: First submitted 2018-03-14; First posted 2018-03-30 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-07

CONDITIONS: Healthy Subjects
Keywords: Drug-alcohol interaction; Lemborexant; E2006; Postural stability; Cognitive performance
MeSH Terms: interventions — lemborexant; Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lemborexant (Experimental): Participants will be randomized to receive a 10 milligram (mg) lemborexant tablet administered with 50 milliliter (mL) water followed by a total volume of 300 mL (approximately 150 mL per aliquot) of a low-calorie beverage (e.g., cranberry beverage) after an overnight fast of at least 8 hours and a sleep period of at least 8 hours. Treatment will be administered after a light breakfast (ie, not high fat), at approximately 120 minutes after wake time in the morning.
  Interventions: Drug: Lemborexant
- Lemborexant Plus Alcohol (Experimental): Participants will be randomized to receive a 10 mg lemborexant tablet administered with 50 mL water followed by alcohol (0.6 grams per kilogram [g/kg] of alcohol for females or 0.7 g/kg of alcohol for males) for a total volume of 300 mL (approximately 150 mL per aliquot) of a low-calorie beverage (e.g., cranberry beverage) after an overnight fast of at least 8 hours and a sleep period of at least 8 hours. Treatment will be administered after a light breakfast (ie, not high fat), at approximately 120 minutes after wake time in the morning.
  Interventions: Drug: Lemborexant; Drug: Alcohol
- Alcohol (Experimental): Participants will be randomized to receive a 10 mg lemborexant-matched placebo tablet administered with 50 mL water followed by alcohol (0.6 g/kg of alcohol for females or 0.7 g/kg of alcohol for males) for a total volume of 300 mL (approximately 150 mL per aliquot) of a low-calorie beverage (e.g., cranberry beverage) after an overnight fast of at least 8 hours and a sleep period of at least 8 hours. Treatment will be administered after a light breakfast (ie, not high fat), at approximately 120 minutes after wake time in the morning.
  Interventions: Drug: Alcohol; Drug: Placebo
- Placebo (Placebo Comparator): Participants will be randomized to receive a 10 mg lemborexant-matched placebo tablet administered with 50 mL water followed by alcohol for a total volume of 300 mL (approximately 150 mL per aliquot) of a low-calorie beverage (e.g., cranberry beverage) after an overnight fast of at least 8 hours and a sleep period of at least 8 hours. Treatment will be administered after a light breakfast (ie, not high fat), at approximately 120 minutes after wake time in the morning.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lemborexant — Film-coated oral tablet
  Arms: Lemborexant; Lemborexant Plus Alcohol
Drug: Alcohol — 0.6 g/kg (female) or 0.7 g/kg (male) of 40% ethanol (volume per volume) vodka diluted in a low-calorie beverage (e.g., cranberry beverage), for a total volume of 300 mL (approximately 150 mL per aliquot).
  Other Names: E2006
  Arms: Alcohol; Lemborexant Plus Alcohol
Drug: Placebo — Film-coated oral tablet
  Arms: Alcohol; Placebo

SUMMARY:
This study will be conducted to evaluate the effects on cognitive performance (Power of Attention domain) and postural stability of lemborexant in combination with alcohol versus lemborexant alone and versus alcohol alone in healthy participants. This study will also assess the safety and tolerability of a single oral dose of lemborexant when administered alone or in combination with alcohol in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be included in this study:

* Healthy male or female, 19 to 55 years of age, inclusive, at the time of informed consent.
* Body mass index ≥22 kilograms per meters squared (kg/m^2) and ≤33 kg/m^2 and a minimum weight of 55.0 kilogram (kg) at Screening
* Current alcohol users who are occasional or regular drinkers, operationally defined as consuming at least 2 alcoholic beverages per week but not more than 2 alcoholic beverages per day in an average week, in the 6 months before Screening. This would result in consumption of 2 to 14 standard drinks per week, on average; 1 standard drink is equivalent to 43 mL (1.5 ounce [oz.]) of spirits (≥20% alcohol by volume), 142 mL (5 oz.) of wine, or 341 mL (12 oz.) of beer.
* Able to speak, read, and understand English sufficiently to allow completion of all study assessments.
* Provide written informed consent.

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from this study:

* Females who are breastfeeding or pregnant.
* Females of childbearing potential. Note: All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
* History of moderate or severe alcohol use disorder within the past 2 years (as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition), and/or participated in, is currently participating in, or is seeking treatment for substance and/or alcohol-related disorders (excluding nicotine and caffeine).
* Presence of insomnia, narcolepsy, obstructive sleep apnea, or restless legs syndrome or an exclusionary score on either of the following subscales of the SLEEP50 questionnaire:

  1. ≥15 on Apnea subscales
  2. ≥7 on Narcolepsy subscale.
* Current or prior diagnosis of any condition for which alcohol consumption is contraindicated (e.g., hypertriglyceridemia, pancreatitis, liver disease, porphyria, or congestive heart failure, judged as clinically relevant by the investigator).
* Evidence of disease that may influence the outcome of the study within 4 weeks prior to the first dose of study drug (e.g., congenital abnormality in metabolism, psychiatric disorders, and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system).
* Has been diagnosed with cancer within the 5 years before Screening (excluding squamous or basal cell carcinoma of the skin), or has an active malignancy of any type (including squamous or basal cell carcinoma of the skin).
* Known history of clinically significant drug allergy at Screening.
* Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening.
* Heavy smokers (≥20 cigarettes per day on average in the past 30 days prior to Screening), chews tobacco, uses a nicotine transdermal patch (including nicotine-containing products) or electronic cigarettes, and/or is unable to abstain from smoking for at least 10 hours during any day.
* Any clinically abnormal symptom or organ impairment found by reviewing medical history at Screening, physical examinations, vital signs, electrocardiogram finding (e.g., a prolonged corrected QT [QTc] interval >450 milliseconds [ms]), or laboratory test results at Screening or Day -1 that require medical treatment or based on the investigator's opinion could affect the safety of the participant.
* Presence of orthostatic hypotension (≥30 millimeter of mercury [mmHg] drop in systolic blood pressure, or ≥20 mmHg drop in diastolic blood pressure) at Screening.
* Any history of gastrointestinal surgery that may affect pharmacokinetic of the study drug (e.g., hepatectomy, digestive organ resection).
* Positive urine drug test at Screening or Day -1; participants positive for tetrahydrocannabinol may be rescheduled at the discretion of the investigator.
* Positive breath alcohol test; participants with positive breath alcohol test may be rescheduled at the discretion of the investigator.
* Weight loss or gain of greater than 10% between Screening and dosing in each Treatment Period. Participants who are currently on, or plan to be on, a restrictive diet will be excluded at the discretion of the investigator.
* Known to be human immunodeficiency virus positive.
* Active viral hepatitis (B or C), as determined by positive serology at Screening.
* Donation or loss of more than 500 mL of whole blood within 30 days preceding the first dose of study drug.
* Treatment with an investigational drug within 28 days or 5-half-lives, whichever is longer, preceding the first dose of study drug. If the half-life is unknown, a 28-day period will apply.
* Use of prescription drugs within 2 weeks prior to dosing.
* Intake of over-the-counter medications within 2 weeks prior to dosing.
* Difficulty with venous access or unsuitable or unwilling to undergo catheter insertion.
* An employee of the sponsor or research site personnel directly affiliated with this study or their immediate family member defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Has current pending legal charges or is currently on probation.
* Unwilling to be searched (including personal effects) for illicit substances before admission to or during the inpatient stays at the research clinic.
* In the opinion of the investigator, is considered unsuitable or unlikely to comply with the study protocol for any reason, including compliance with the study prohibitions and restrictions and completion of the cognitive performance and postural stability tasks.
* Previously participated in any clinical trial of lemborexant.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in body sway, as assessed by an ataxia meter measuring directional trunk movements, for lemborexant plus alcohol compared to lemborexant alone | Baseline; Up to approximately 12 weeks postdose in each single-dose treatment period
  Body sway will be detected through a cable around the participant's waist by the ataxia meter. Body sway will be measured in units of 1/3° of the angle of arc. For ease in reporting, these will be called arbitrary units, with a higher number indicating more body sway (less postural stability).
Change from baseline in body sway, as assessed by an ataxia meter measuring directional trunk movements, for lemborexant plus alcohol compared to alcohol alone | Baseline; Up to approximately 12 weeks postdose in each single-dose treatment period
  Body sway will be detected through a cable around the participant's waist by the ataxia meter. Body sway will be measured in units of 1/3° of the angle of arc. For ease in reporting, these will be called arbitrary units, with a higher number indicating more body sway (less postural stability).
Change from baseline in Power of Attention, per the Performance Assessment Battery (PAB), for lemborexant plus alcohol compared to lemborexant alone | Baseline; Up to approximately 12 weeks postdose in each single-dose treatment period
  The PAB comprises 9 tasks: Simple Reaction Time; Choice Reaction Time; Digit Vigilance; Immediate Word Recall; Delayed Word Recall; Numerical Working Memory; Spatial Working Memory; Word Recognition; Picture Recognition. Four composite domain factor scores will be calculated by combining outcome variables from the various tests. The 4 domains are Power of Attention, Continuity of Attention, Quality of Memory, and Speed of Memory Retrieval. The Power of Attention score is a composite score from the speed scores of 3 tests of attention (Simple Reaction Time, Choice Reaction Time, Digit Vigilance) and reflects the ability to focus attention and process information. A higher score indicates better performance.
Change from baseline in Power of Attention, per the PAB, for lemborexant plus alcohol compared to alcohol alone | Baseline; Up to approximately 12 weeks postdose in each single-dose treatment period
  The PAB comprises 9 tasks: Simple Reaction Time; Choice Reaction Time; Digit Vigilance; Immediate Word Recall; Delayed Word Recall; Numerical Working Memory; Spatial Working Memory; Word Recognition; Picture Recognition. Four composite domain factor scores will be calculated by combining outcome variables from the various tests. The 4 domains are Power of Attention, Continuity of Attention, Quality of Memory, and Speed of Memory Retrieval. The Power of Attention score is a composite score from the speed scores of 3 tests of attention (Simple Reaction Time, Choice Reaction Time, Digit Vigilance) and reflects the ability to focus attention and process information. A higher score indicates better performance.

SECONDARY OUTCOMES:
Mean value of maximum observed concentration (Cmax) for lemborexant and its metabolites (M4, M9, and M10) | Predose; 0.5, 1.5, 2, 3, 4, 6, 9, 12, 24, 36, 48, and 72 hours postdose in each single-dose treatment period
  Blood samples will be collected for the determination of plasma Cmax.
Mean value of time at which the maximum drug concentration is observed (tmax) for lemborexant and its metabolites (M4, M9, and M10) | Predose; 0.5, 1.5, 2, 3, 4, 6, 9, 12, 24, 36, 48, and 72 hours postdose in each single-dose treatment period
  Blood samples will be collected for the determination of plasma tmax.
Mean value of area under the concentration-time curve from zero time to time of last quantifiable concentration (AUC0-t) for lemborexant and its metabolites (M4, M9, and M10) | Predose; 0.5, 1.5, 2, 3, 4, 6, 9, 12, 24, 36, 48, and 72 hours postdose in each single-dose treatment period
  Blood samples will be collected for the determination of plasma AUC0-t.
Mean value of area under the concentration-time curve from zero time to 9 hours after dosing (AUC0-9h) for lemborexant | Predose; 0.5, 1.5, 2, 3, 4, 6 and 9 hours postdose in each single-dose treatment period
  Blood samples will be collected for the determination of plasma AUC0-9h.
Mean value of area under the concentration-time curve from zero time to 12 hours after dosing (AUC0-12h) for lemborexant and its metabolites (M4, M9, and M10) | Predose; 0.5, 1.5, 2, 3, 4, 6, 9 and 12 hours postdose in each single-dose treatment period
  Blood samples will be collected for the determination of plasma AUC0-12h.
Mean value of area under the concentration-time curve from zero time to 24 hours after dosing (AUC0-24h) for lemborexant and its metabolites (M4, M9, and M10) | Predose; 0.5, 1.5, 2, 3, 4, 6, 9, 12 and 24 hours postdose in each single-dose treatment period
  Blood samples will be collected for the determination of plasma AUC0-24h.
Mean value of area under the concentration-time curve from zero time to 48 hours after dosing (AUC0-48h) for lemborexant and its metabolites (M4, M9, and M10) | Predose; 0.5, 1.5, 2, 3, 4, 6, 9, 12, 24, 36 and 48 hours postdose in each single-dose treatment period
  Blood samples will be collected for the determination of plasma AUC0-48h.
Mean value of area under the concentration-time curve from zero time to 72 hours after dosing (AUC0-72h) for lemborexant and its metabolites (M4, M9, and M10) | Predose; 0.5, 1.5, 2, 3, 4, 6, 9, 12, 24, 36, 48, and 72 hours postdose in each single-dose treatment period
  Blood samples will be collected for the determination of plasma AUC0-72h.
Mean value of terminal elimination phase half-life (t1/2) for lemborexant and its metabolites (M4, M9, and M10) | Predose; 0.5, 1.5, 2, 3, 4, 6, 9, 12, 24, 36, 48, and 72 hours postdose in each single-dose treatment period
  Blood samples will be collected for the determination of plasma t1/2.
Mean value of apparent total body clearance (CL/F) for lemborexant after extravascular administration | Predose; 0.5, 1.5, 2, 3, 4, 6, 9, 12, 24, 36, 48, and 72 hours postdose in each single-dose treatment period
  Blood samples will be collected for the determination of plasma CL/F.
Mean value of AUC0-9h after dosing, metabolite ratio for lemborexant and its metabolites (M4, M9, and M10) | Predose; 0.5, 1.5, 2, 3, 4, 6 and 9 hours postdose in each single-dose treatment period
  The metabolite ratio is defined as the ratio of lemborexant metabolite to lemborexant AUC0-9h, corrected for molecular weight. Blood samples will be collected for the determination of plasma AUC0-9h.
Mean value of AUC0-12h after dosing, metabolite ratio for lemborexant and its metabolites (M4, M9, and M10) | Predose; 0.5, 1.5, 2, 3, 4, 6, 9 and 12 hours postdose in each single-dose treatment period
  The metabolite ratio is defined as the ratio of lemborexant metabolite to lemborexant AUC0-12h, corrected for molecular weight. Blood samples will be collected for the determination of plasma AUC0-12h.
Mean value of AUC0-24h after dosing, metabolite ratio for lemborexant and its metabolites (M4, M9, and M10) | Predose; 0.5,1.5, 2, 3, 4, 6, 9,12 and 24 hours postdose in each single-dose treatment period
  The metabolite ratio is defined as the ratio of lemborexant metabolite to lemborexant AUC0-24h, corrected for molecular weight. Blood samples will be collected for the determination of plasma AUC0-24h.
Mean AUC0-48h after dosing, metabolite ratio for lemborexant and its metabolites (M4, M9, and M10) | Predose; 0.5, 1.5, 2, 3, 4, 6, 9, 12, 24, 36 and 48 hours postdose in each single-dose treatment period
  The metabolite ratio is defined as the ratio of lemborexant metabolite to lemborexant AUC0-48h, corrected for molecular weight. Blood samples will be collected for the determination of plasma AUC0-48h.
Mean value AUC0-72h after dosing, metabolite ratio for lemborexant and its metabolites (M4, M9, and M10) | Predose; 0.5, 1.5, 2, 3, 4, 6, 9, 12, 24, 36, 48, and 72 hours postdose in each single-dose treatment period
  The metabolite ratio is defined as the ratio of lemborexant metabolite to lemborexant AUC0-72h, corrected for molecular weight. Blood samples will be collected for the determination of plasma AUC0-72h.
Mean value of time interval from dosing to the first measureable concentration (tlag) for lemborexant and its metabolites (M4, M9, and M10) | Predose; 0.5, 1.5, 2, 3, 4, 6, 9, 12, 24, 36, 48, and 72 hours postdose in each single-dose treatment period
  Blood samples will be collected for the determination of plasma tlag.
Change from baseline in Continuity of Attention, per the PAB, for lemborexant plus alcohol compared to lemborexant alone, lemborexant plus alcohol compared to alcohol alone, and alcohol compared to placebo | Baseline; Up to approximately 12 weeks postdose in each single-dose treatment period
  The PAB is comprised of 9 tasks: Simple Reaction Time; Choice Reaction Time; Digit Vigilance; Immediate Word Recall; Delayed Word Recall; Numerical Working Memory; Spatial Working Memory; Word Recognition; Picture Recognition. Four composite domain factor scores will be calculated by combining outcome variables from the various tests. The 4 domains are Power of Attention, Continuity of Attention, Quality of Memory, and Speed of Memory Retrieval. The Continuity of Attention score is a composite score created by combining the accuracy scores from the 3 tests of attention (Simple Reaction Time, Choice Reaction Time, Digit Vigilance) and reflects the ability to sustain attention (vigilance). A higher score indicates better performance.
Change from baseline in Quality of Memory, per the PAB, for lemborexant plus alcohol compared to lemborexant alone, lemborexant plus alcohol compared to alcohol alone, and alcohol compared to placebo | Baseline; Up to approximately 12 weeks postdose in each single-dose treatment period
  The PAB is comprised of 9 tasks: Simple Reaction Time; Choice Reaction Time; Digit Vigilance; Immediate Word Recall; Delayed Word Recall; Numerical Working Memory; Spatial Working Memory; Word Recognition; Picture Recognition. Four composite domain factor scores will be calculated by combining outcome variables from the various tests. The 4 domains are Power of Attention, Continuity of Attention, Quality of Memory, and Speed of Memory Retrieval. The Quality of Memory score is a composite score created by combining the accuracy measures from the 2 tests of working memory and the 4 tests of episodic memory (Numeric Working Memory, Spatial Working Memory, Immediate Word Recall, Delayed Word Recall, Word Recognition, Picture Recognition) and reflects the ability to store information in memory and subsequently retrieve it. A higher score indicates better performance.
Change from baseline in Speed of Memory Retrieval, per the PAB, for lemborexant plus alcohol compared to lemborexant alone, lemborexant plus alcohol compared to alcohol alone, and alcohol compared to placebo | Baseline; Up to approximately 12 weeks postdose in each single-dose treatment period
  The PAB is comprised of 9 tasks: Simple Reaction Time; Choice Reaction Time; Digit Vigilance; Immediate Word Recall; Delayed Word Recall; Numerical Working Memory; Spatial Working Memory; Word Recognition; Picture Recognition. Four composite domain factor scores will be calculated by combining outcome variables from the various tests. The 4 domains are Power of Attention, Continuity of Attention, Quality of Memory, and Speed of Memory Retrieval. The Speed of Memory Retrieval score is a composite score created by combining the reaction time scores from the 2 working memory tests and the 2 episodic recognition tests (Numeric Working Memory, Spatial Working Memory, Word Recognition, Picture Recognition) and reflects time taken to retrieve information held in both working and episodic memory. A higher score indicates better performance.
Change from baseline in body sway, as assessed by an ataxia meter measuring directional trunk movements, for alcohol compared to placebo | Baseline; Up to approximately 12 weeks postdose in each single-dose treatment period
  Body sway will be detected through a cable around the participant's waist by the ataxia meter. Body sway will be measured in units of 1/3° of the angle of arc. For ease in reporting, these will be called arbitrary units, with a higher number indicating more body sway (less postural stability).
Change from baseline in Power of Attention, per the PAB, for alcohol compared to placebo | Baseline; Up to approximately 12 weeks postdose in each single-dose treatment period
  The PAB is comprised of 9 tasks: Simple Reaction Time; Choice Reaction Time; Digit Vigilance; Immediate Word Recall; Delayed Word Recall; Numerical Working Memory; Spatial Working Memory; Word Recognition; Picture Recognition. Four composite domain factor scores will be calculated by combining outcome variables from the various tests. The 4 domains are Power of Attention, Continuity of Attention, Quality of Memory, and Speed of Memory Retrieval. The Power of Attention score is a composite score from the speed scores of 3 tests of attention (Simple Reaction Time, Choice Reaction Time, Digit Vigilance) and reflects the ability to focus attention and process information. A higher score indicates better performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health, Toronto, Ontario, Canada